CLINICAL TRIAL: NCT05968547
Title: Evaluation of Patients' Requirements for Improved Advice and Guidance on Vision Standards for Driving in Glaucoma
Acronym: D&G
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B00964
Record Dates: First submitted 2023-07-19; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Glaucoma
Keywords: Driving Standards; DVLA; Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Glaucoma patients questionnaire: Questionnaire to understand patients driving needs and understanding of driving vision standards
- Visual acuity standards: DVLA vision standard estimated in the clinic is compared with standandard car number plate outside the clinic. We estimate the vision in the clinic using standard visual acuity chart and electronic number plate vision and compare with number plate vision estimated outside the clinic by the patient. Instruction to estimate number plate vision will be provided to the patient.
  Interventions: Other: Driving assessment in glaucoma patient

INTERVENTIONS:
Other: Driving assessment in glaucoma patient — One group of patient will be given questionnaire while the other group will respond to a questionnaire while the other group will have vision assessment. Patients could participate in both groups.
  Other Names: 1. questionnaire to patient. 2.Assessment of vision using visual acuity chart and number plate vision
  Groups: Visual acuity standards

SUMMARY:
Glaucoma can affect both central and peripheral vision. Clinicians need to discuss with patients the vision related driving standards and any specific limitations their patients may have relating to their ability to drive with glaucoma. According to the recent guidelines by the General Optical Council (GOC), clinicians are advised to make sure that the Driving and Vehicle Licensing Agency (DVLA) is informed about patients who do not meet the driving vision standards. There are several limitations in making a professional judgement about a patient's suitability to drive and in providing appropriate advice to patients. The main concern is discussing this sensitive issue with the patient based upon available clinical evidence e.g. vision or visual field and directing them to inform the DVLA of their condition or potentially advising them to stop driving. The purpose of this research is to investigate the two main issues 1. To explore patients' understanding of standards of vision for driving. 2. Comparing the standards of vision for driving estimated in the clinic with number plate vision. We propose to do a mixed methods analysis using a patient survey and quantitative investigation of driving vision standards.

DETAILED DESCRIPTION:
The two main objectives that we propose to study in this project are

1. Descriptive understanding of patients' perception of their driving needs and their understanding of driving standards. This will be studied with the help of a survey questionnaire to learn about patients' driving needs, sight history, understanding of DVLA vision standards and the driving advice given to them. Understanding glaucoma patients' general perceptions about standards of vision for driving and their driving needs will help us to improve communication with the patients and to give the best possible advice about standards of vision for driving.
2. Quantitative comparison of standards of vision for driving as required by DVLA and clinical vision assessment in glaucoma patients. The limitations to meet the vision standard for driving will be assessed in glaucoma patients in the clinic and outside the clinic as required by DVLA standards of vision for driving. In the clinic, vision will be assessed by checking if the patient can binocularly read the 6/12 line on the vision chart and electronic number plate test used in the clinic. The results will be compared with a self-assessed number plate vision - a standard requirement to meet DVLA's standard of vision for driving. Understanding the clinical estimation of binocular vision, patients' ability to read the number plate in clinic and to self-assess their number plate vision will help the clinician to know patients' abilities and give evidence-based advice to the glaucoma patient about meeting the DVLA standards of vision.

ELIGIBILITY:
Inclusion criteria for Patient survey:

* All patients attending the glaucoma clinic will be eligible for the survey.
* Both drivers and non-drivers will be included in the study.

Inclusion Criteria for Quantitative vision estimation:

• Glaucoma patients with habitual vision of 6/19 or better at least in one eye (whether driving or not driving).

Exclusion criteria for Patient survey:

• All the patients attending glaucoma clinic, willing to participate in the study, will be eligible to participate in the survey and will not be excluded from the study.

Exclusion Criteria for Quantitative vision estimation:

• Patients with a binocular habitual visual acuity of less than 6/19 will not be able to eligible to participate in qualitative vision assessment.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending glaucoma clinics.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-25 (Estimated); Primary Completion 2023-10-25 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Ability to read 6/12 or above in vision chart with both eyes. | 6 months
  Binocular Vision assessment in Logmar testing
Vision Chart score in each eye | 6 months
  Unilateral Vision testing Logmar testing
Ability to read the number plate in the clinic displayed in the VDU | 6 months
  Ability to read the number plate in the clinic displayed in the VDU comparative visual display unit
Ability to read the car number plate outside the clinic | 6 months
  Ability to read the car number plate outside the clinic as per patients self assessment

CONTACTS AND LOCATIONS:
Overall Officials: Subash Sukumar, Principal Investigator — Manchester Royal Eye Hospital
Locations (1):
- Manchester Royal Eye Hospital, Manchester, United Kingdom